CLINICAL TRIAL: NCT00909025
Title: Clinical First-in-human Single-dose Escalation Study Evaluating the Safety and Tolerability of Claudiximab (iMAB-362) in Hospitalized Patients With Advanced Gastroesophageal Cancer. A Multi-center, Phase I, Open-label, i.v. Infusion Study
Brief Title: Safety and Tolerability Study of Claudiximab in Patients With Advanced Gastroesophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ganymed Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GM-IMAB-001
Record Dates: First submitted 2009-05-18; First posted 2009-05-27 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumors
MeSH Terms: interventions — zolbetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Claudiximab (Experimental)
  Interventions: Drug: Claudiximab

INTERVENTIONS:
Drug: Claudiximab — Patients receive Claudiximab as intravenous infusion over 2 hours on day 1. Cohorts of 3-6 patients receive escalating doses of Claudiximab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no dose-limiting toxicity (DLT) is diagnosed in 3 patients or no more than 1 out of 6 patients exhibits a DLT.
  After completion of study treatment, patients are followed for 4 weeks.

SUMMARY:
Claudiximab is a monoclonal antibody specific for gastric and gastroesophageal adenocarcinomas. Preclinically, claudiximab was shown to inhibit tumor growth and to kill cancer cells by indirect (complement-dependent cytoxicity, antibody-dependent cellular cytotoxicity) and direct mechanisms (antiproliferative and proapoptotic effects). The aim of this phase I study is to establish safety, toxicity and maximal tolerable dose of a single infusion of claudiximab in patients suffering from relapsing, advanced gastroesophageal and gastric adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* Metastatic, refractory or recurrent disease of advanced gastroesophageal cancer (adenocarcinoma) proven by histology
* CLDN18.2 expression confirmed by immunohistochemistry
* Prior standard chemotherapy containing a fluoropyrimidine, a platinum compound and/or epirubicine, and - if clinically appropriate - docetaxel
* At least 1 measurable site of the disease according RECIST criteria (CT-scans or MRT not older than 6 weeks before study entry)
* Age ≥ 18 years
* ECOG performance status (PS) 0-1 or Karnofsky Index 70-100%
* Life expectancy > 3 months
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dl
* INR < 1.5
* Bilirubin normal
* AST and ALT < 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Creatinine < 1.5 x ULN

Exclusion Criteria:

* Pregnancy or breastfeeding
* Prior allergic reaction or intolerance to a monoclonal antibody
* Prior inclusion in the present study
* Less than 3 weeks since prior anti-tumor or radiation therapy
* Other investigational agents or devices concurrently or within 4 weeks prior to this study
* Other concurrent anticancer therapies
* History of positive test for human immunodeficiency virus (HIV) antibody
* Known Hepatitis.
* Uncontrolled or severe illness.
* Concurrent administration of anticoagulation agents with vitamin K antagonists
* Concurrent administration of therapeutic doses of heparin (prophylactic doses are acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-05-31 (Actual); Primary Completion 2010-05-31 (Actual); Study Completion 2010-05-31 (Actual)

PRIMARY OUTCOMES:
Determination of maximum tolerated dose of claudiximab (Phase I: toxicities as assessed by NCI CTCAE version 3.0) | Four weeks

SECONDARY OUTCOMES:
Determination of the safety profile | Four weeks
Pharmacokinetic evaluation | Four weeks
Overall tumor response as assessed by RECIST | Four weeks
Evaluation of immunogenicity | Four weeks
Determination of antitumoral efficacy | Four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schuler, Prof.Dr.med., Principal Investigator — Innere Klinik (Tumorforschung) Universitätsklinikum Essen Hufelandstr. 55 45122 Essen, GERMANY
Locations (6):
- Germany (4):
  - Universitätsklinikum Essen, Innere Klinik (Tumorforschung), Essen
  - Universität Heidelberg, Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
  - Johannes Gutenberg Universität, 1.Med Klinik und Poliklinik, Mainz
  - Klinikum Rechts-der-Isar, III.Medizinische Klinik und Poliklinik, München
- Latvia (2):
  - Piejuras Hospital, Liepāja
  - Pauls Stradins University, Riga

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Sahin U, Schuler M, Richly H, Bauer S, Krilova A, Dechow T, Jerling M, Utsch M, Rohde C, Dhaene K, Huber C, Tureci O. A phase I dose-escalation study of IMAB362 (Zolbetuximab) in patients with advanced gastric and gastro-oesophageal junction cancer. Eur J Cancer. 2018 Sep;100:17-26. doi: 10.1016/j.ejca.2018.05.007. Epub 2018 Jun 21. PMID 29936063
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website — https://www.clinicaltrials.astellas.com/study/GM-IMAB-001/
- See also: Link to plain language summary of the study on the Trial Results Summaries website — https://www.trialsummaries.com/Study/StudyDetails?id=25770&tenant=MT_AST_9011